CLINICAL TRIAL: NCT04769141
Title: Artificial Intelligence Guided Personalised Medicine in Patients With Hypertension and Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alexandra Hospital (Other)
Responsible Party: Principal Investigator, Amartya Mukhopadhyay, Senior Consultant, Division of Respiratory & Critical Care Medicine, Department of Medicine, National University Hospital, Alexandra Hospital
Other Study IDs: AlexandraHosp
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension patients: a prospective 4-month, cohort feasibility study will evaluate blood pressure (n=20) using the CURATE.AI platform.
  Interventions: Combination Product: CURATE.AI
- Diabetic patients: a prospective 4-month, cohort feasibility study will evaluate glycaemic (n=20) control using the CURATE.AI platform.
  Interventions: Combination Product: CURATE.AI

INTERVENTIONS:
Combination Product: CURATE.AI — CURATE.AI is one example of an artificial intelligence guided dosing decision tool. It is customized to each individual and can be applicable across many different conditions, as it is disease agnostic.
  This platform has already demonstrated initial success in cancer and transplant populations but yet to be applied to chronic disease patients.

SUMMARY:
Hypertension and diabetes are chronic diseases that require long-term management and disease control is often sub-optimal, leading to complications which place additional burden on patients and the healthcare system.

This study aims to address factors such as gender, ethnicity and specific genetics that are not routinely considered during drug dosing but account for considerable variations in drug responses by tailoring the treatment to individual patient using CURATE.AI. CURATE.AI is an artificial intelligence guided dosing decision tool and can be applicable across many different conditions, as it is disease agnostic. This platform had demonstrated initial success in cancer and transplant populations but has yet to be applied to chronic disease patients.

The aim of this study is demonstrate that artificial intelligence guided treatment in chronic disease of hypertension and type 2 diabetes mellitus will yield actionable medication dosing optimization.

DETAILED DESCRIPTION:
The aim of this study is demonstrate that artificial intelligence guided treatment in chronic disease of hypertension and type 2 diabetes mellitus will yield actionable medication dosing optimization.

Study Objectives

1. Artificial intelligence (CURATE.AI) pilot deployment using prospective data in patients with hypertension and type 2 diabetes mellitus.
2. Artificial intelligence (CURATE.AI) for behavioural assessment and compliance prediction to disease management programme in patients with hypertension and type 2 diabetes mellitus.

Methods and Analysis Design and setting

This prospective cohort feasibility study will evaluate the blood pressure (n=20) and glycaemic (n=20) control of patients using the CURATE.AI platform. Participants will be recruited for a period of 4 months from the day of baseline visit and followed up for up to 4 clinic visits.

Recruitment Participants will be recruited from the study site, Alexandra Hospital, Singapore during their routine clinic visits. The doctor will identify individuals who meet the inclusion criteria and the research team will share further details regarding the study including the inclusion/ exclusion criteria that is presented below.

Interested individuals who meet the eligibility criteria will be required to sign the Informed Consent From prior to any study activity and a baseline visit will be scheduled.

Inclusion criteria

* Adult patients (≥ 21years) with T2DM or hypertension
* Expected to be followed up in Alexandra Hospital for the next 4-months
* Signed informed consent form

Exclusion criteria

* Patients with cognitive impairment
* Patients with active cancer undergoing chemotherapy
* Patients on haemodialysis or peritoneal dialysis (which can cause rapid fluctuation of BP and blood sugar, respectively)
* Pregnant patients
* Patients whose medications for T2DM and hypertension are changed simultaneously during the first clinic visit
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.

Study procedures The CURATE.AI correlation requires three data-points to calculate the initial drug dose. Ongoing readings provide further data-points for dose modulation.

Once a patient with hypertension or T2DM is identified and consented, a BP or blood sugar will be recorded (1st data-point) and baseline assessment performed

Following any change of hypertension (or T2DM) medications, a 24-hour ambulatory BP (or continuous glucose monitoring) will be done during the 7-15 days after baseline visit (data-point 2 or data-point 3 if retrospective data is available). Data from these recordings will be used to titrate medications, if necessary, in the follow-up visits.

One month after baseline the patient will return to the clinic for follow-up (data-point 3 or data point 4 if retrospective data is available) and dose adjustment, if required.

Dosing decisions at this point and going forward will be made by CURATE.AI and verified by the clinician. If dose adjustment is required, then the patient will repeat the home monitoring (24-hour ambulatory BP or continuous glucose monitoring). If dose adjustment is not needed the patient will undertake no home monitoring. Either way each patient will return one month later for clinic follow-up (clinic visit 2). This monthly cycle is repeated until each patient has reached 4-months follow-up.

At the final clinic visit (4-months after baseline) the baseline assessments are repeated. At this point patients will also be approached to complete a patient experience survey.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 21years) with T2DM or hypertension
* Expected to be followed up in Alexandra Hospital for the next 4-months
* Signed informed consent form

Exclusion Criteria:

* Patients with cognitive impairment
* Patients with active cancer undergoing chemotherapy
* Patients on hemodialysis or peritoneal dialysis (which can cause rapid fluctuation of BP and blood sugar, respectively)
* Pregnant patients
* Patients whose medications for T2DM and hypertension are changed simultaneously during the first clinic visit
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with a clinically confirmed diagnosis of T2DM and 20 patients with a diagnosis of hypertension will be screened, recruited and followed up.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Medication dosing optimization | 3 years
  • Artificial intelligence guided treatment in chronic disease of hypertension and type 2 diabetes mellitus will yield actionable medication dosing optimization and to demonstrate technical development of artificial intelligence platform (CURATE.AI) using retrospective data in patients with hypertension and type 2 diabetes mellitus.

SECONDARY OUTCOMES:
(CURATE.AI) pilot deployment using prospective data | 3 years
  • Artificial intelligence (CURATE.AI) for behavioural assessment and compliance prediction to disease management programme in patients with hypertension and type 2 diabetes mellitus.

IPD SHARING:
Plan to Share IPD: Undecided